CLINICAL TRIAL: NCT03327259
Title: A Pilot Study of Therapist Guided Activity Practice for Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Aliza T. Stein, Doctoral Student, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-02-0043
Record Dates: First submitted 2017-10-23; First posted 2017-10-31 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression | interventions — Ambulatory Care Facilities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity Planning Only (Active Comparator)
  Interventions: Behavioral: Activity Planning
- Enhanced Activity Planning (Experimental): Activity planning with therapist guided activity practice.
  Interventions: Behavioral: Activity Planning; Behavioral: Therapist Guided Activity Practice

INTERVENTIONS:
Behavioral: Activity Planning — The therapist will work with the participant to select a challenging, yet rewarding or value-driven activity that he/she can engage in 5x and monitor daily over the upcoming week.
Behavioral: Therapist Guided Activity Practice — The therapist will work with the participant to plan and carry out a brief in-vivo version of their goal/target activity. The therapist will guide the participant through the activity for approximately 15 minutes.
  Arms: Enhanced Activity Planning

SUMMARY:
There is literature to support both the need for and efficacy of brief interventions for depressive symptoms, particularly among college students.Brief behavioral activation interventions (BATD) have gained recognition as efficacious treatments for depression; yet a recent study evidenced a substantial (39%) non-response rate (Kuyken et al., 2017). In accordance with behavioral models of depression, the treatment involves increasing activity and positive experience, to break the negative reinforcement cycle maintaining depressed mood. Thus, strategies that may facilitate increasing activity may improve BATD outcomes. The objective of the current study is to examine whether briefly practicing a target activity during an activity planning session (modified single session of BATD) increases the likelihood of completing the activity during the upcoming week. We hypothesized that guided activity practice may improve self-efficacy within session and activity completion in the upcoming week. We further aim to explore whether activity completion mediates depressive symptom change.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* University of Texas at Austin students currently enrolled in Introductory Psychology (PSY 301)
* Score >14 on Beck Depression Inventory during both pre-screening and baseline screen
* Avoidance rating >59 and Distress rating >39 on at least one item of the Avoidance Screen.

Exclusion Criteria:

* Initiated psychotherapy or psychotropic medication in past 6 weeks
* Recent change (past 6 weeks) in psychotropic medication
* Current or past psychosis or mania

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Percent Activity Completion Between Conditions | Daily for 7 days
  Participants will complete daily surveys for seven days following the initial visit. Participants will answer whether or not the activity was completed that day. Data will be collected using Qualtrics survey software. The outcome variable is the percentage of days the participant completed the activity.
Change in Self-Efficacy in Response to Therapist Guided Activity Practice | Baseline
  Following the activity planning portion of the initial visit, participants rate the degree of self-efficacy (confidence in ability to complete the goal) on a scale from 0 (no confidence) to 100 (complete confidence). Participants randomized to Enhanced Activity Practice condition will complete a second rating following the activity practice. The pre-to-post difference score in self-efficacy will be examined as a primary outcome.

SECONDARY OUTCOMES:
Depressive Symptoms | Baseline and 1 week follow-up
  Severity of depressive symptoms will be measured at baseline and 1-week follow-up using the Beck Depression Inventory-II.
Experiential Avoidance and Psychological Flexibility | Baseline and 1 week follow-up
  Experiential avoidance and psychological flexibility will be measured at baseline and 1-week follow-up using the Acceptance and Action Questionnaire-II.
Multidimensional Experiential Avoidance | Baseline and 1 week follow-up
  Multidimensional experiential avoidance will be measured at baseline and 1-week follow-up using the Multidimensional Experiential Avoidance Questionnaire.

OTHER OUTCOMES:
Behavioral Activation | Baseline and 1 week follow-up
  Behavioral Activation will be measured at baseline and 1-week follow-up using the Behavioral Activation for Depression Scale.
Distress Intolerance | Baseline and 1 week follow-up
  Distress intolerance will be measured at baseline and 1-week follow-up using the Distress Intolerance Index.
Anxiety Sensitivity and Distress Intolerance | Baseline and 1 week follow-up
  As an additional measure of distress intolerance, the Anxiety Sensitivity Index will be measured at baseline and 1-week follow-up.
Anxiety Symptoms | Baseline and 1 week follow-up
  Anxiety symptoms will be measured at baseline and 1-week follow-up using the Beck Anxiety Inventory.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided